CLINICAL TRIAL: NCT04030156
Title: ASSESSMENT OF TONSIL VOLUME WITH TRANSCERVICAL ULTRASONOGRAPHY IN BOTH CHILDREN AND ADULTS - A PROSPECTIVE CLINICAL RESEARCH
Brief Title: ASSESMENT OF TONSIL VOLUME WITH ULTRASONOGRAPHY IN BOTH CHILDREN AND ADULTS
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erdem Mengi, Assistant Professor of Otorhinolaryngology, Pamukkale University
Other Study IDs: 60116787-020/56040
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: OSAS; Recurrent Tonsillitis
Keywords: Size; tonsil; tonsillectomy; ultrasonography
MeSH Terms: conditions — Tonsillitis | interventions — Tonsillectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ultrasonographic tonsil volume: All measurements were done by the same radiologist with over 20 years of experience. GE LOGIQ E9 (GE Healthcare, Milwaukee, WI, USA) was used in USG examination. The patients were viewed using a 2-9 MHz linear probe from the submental region. The examination was done while the patient was in a supine position, with a neck support. Right tonsil measurement was done by turning the neck slightly to the upper left whereas left tonsil measurement was done by turning the neck slightly to the upper right. Tonsil volume was calculated with standard ultrasonography formula (height x length x thickness x 0.52) due to its ellipsoid shape.
  Interventions: Procedure: tonsillectomy
- Actual tonsil volume: Excised tonsil volumes were calculated by water replacement method.
  Interventions: Procedure: tonsillectomy

INTERVENTIONS:
Procedure: tonsillectomy — Tonsillectomy was performed under general anesthesia using cold dissection method.

SUMMARY:
The tonsil volume is an important factor in the decision of the tonsillectomy operation. For this reason, it is important to evaluate the tonsil size before the surgery. Ultrasonography was used in a limited number of studies about tonsil tissue assessment and also those studies include only the pediatric population. In this study, we investigate the success of ultrasonography in adults additionally pediatric population as a contribution to literature.

DETAILED DESCRIPTION:
Tonsillectomy is a common procedure performed on both adults and children. Recurrent tonsillitis, snoring and obstructive sleep apnea is among the most important indications for this surgery. Tonsil volume, in addition to recurrent tonsillitis frequency, are both considered in deciding tonsillectomy operation. Moreover, recent studies showed a correlation between tonsil hypertrophy and tonsillitis frequency. For this reason, a reliable assessment of tonsil volume is crucial both during clinical follow-up and surgery decision.

Today, a number of clinical staging systems are used to assess tonsil volume; with 'Friedman Scale' and 'Brodsky Scale' being the most commonly used systems. Those staging systems employ physical examination and are graded on palatine tonsils' midline extension. In other words, clinical staging uses just the transverse length of tonsils and vertical length and depth are dismissed. In addition, other factors such as patient non-compliance, size of the tongue and tongue base, hyperactive gag reflex and trismus make a clinical assessment difficult. For those reasons, a correct clinical assessment of tonsil volume is not always conceivable.

Ultrasonography (USG) was used in a limited number of studies about tonsil tissue assessment despite high patient compliance, low cost and its non-radioactive nature. Also, those studies include only the pediatric population.In this study, we would like to assess the success of USG in objective measurement of tonsil volume in both pediatric and adult populations and comparison of those results with clinical findings

ELIGIBILITY:
Inclusion Criteria:

* Tonsillectomy patients with recurrent tonsillitis
* Tonsillectomy patients with obstructive sleep apnea syndrome.

Exclusion Criteria:

-Tonsillectomy patients with suspected malignancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Both adult and pediatric populations with tonsillectomy indication and diagnosed with recurrent tonsillitis and obstructive sleep apnea syndrome were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical tonsil grade | 20 minutes
  Physical examination of patients and tonsil grade assessment using Friedman tonsil grading system were done prior to surgery
mean ultrasonographic tonsil volume (ml) | 20 minutes
  Tonsil volume was calculated with standard ultrasonography formula (height x length x thickness x 0.52) due to its ellipsoid shape
mean actual tonsil volume (ml) | 20 minutes
  Excised tonsil volumes were calculated by water replacement method.

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Mengi, Principal Investigator — Pamukkale University School of Medicine, Denizli, Turkey
Locations (1):
- Erdem Mengi, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No